CLINICAL TRIAL: NCT05200585
Title: Pilot of Lifestyle Behavior Intervention for Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Principal Investigator, Natalia Heredia, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-21-1008
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Liver/Hígado Sano program (Experimental)
  Interventions: Behavioral: Healthy Liver/Hígado Sano program
- Control Group (Active Comparator)
  Interventions: Behavioral: Usual standard of care

INTERVENTIONS:
Behavioral: Healthy Liver/Hígado Sano program — The program will last 4-6 months and include 16 sessions, each 30-60 minutes long, that focus on self-management strategies for dietary changes and physical activity and is meant to be delivered in 4-6 months. The 16 sessions are as follows: 1) Introduction to the program, 2) Get Active, 3) Track Your Activity, 4) Eat Well, 5) Track Your Food, 6) Get More Active, 7) Burn More Calories Than You Take In, 8) Shop and Cook, 9) Manage Stress, 10) Find Time for Fitness, 11) Cope with Triggers, 12) Keep Your Heart Healthy, 13) Take Charge of Your Thoughts, 14) Get Support, 15) Eat Well Away from Home, and 16) Staying Motivated
  Arms: Healthy Liver/Hígado Sano program
Behavioral: Usual standard of care — Participants will receive ongoing monitoring of condition at the clinic per standard of care and a short informational pamphlet
  Arms: Control Group

SUMMARY:
The purpose of this study is to pilot test a behavioral lifestyle intervention for Hispanic/Latino patients with non-alcoholic fatty liver disease (NAFLD)

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic/Latino
* Have been diagnosed with NAFLD
* Able to speak English or Spanish
* Have access to internet, either on their phone, at home or at some other location convenient to the participant

Exclusion Criteria:

* Does not have a working telephone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited | end of study(6 months after enrollment)
Number of participants that adhere to the intervention | end of study(6 months after enrollment)
Number of participants that complete the study | end of study(6 months after enrollment)
Intervention group participants Satisfaction of program as assessed by the Client Satisfaction Questionnaire (CSQ-8) | end of study(6 months after enrollment)
  The Client Satisfaction Questionnaire (CSQ) has 8 items.Each one is scored from 1-4, with a total possible score of 32, a higher score indicating greater satisfaction

SECONDARY OUTCOMES:
Height of participants | Baseline, 6 months after enrollment
Change in weight of participants | Baseline, 6 months after enrollment
Change in liver function as assessed by alanine aminotransferase (ALT) levels | Baseline, 6 months after enrollment
  Higher levels of ALT indicates liver damage
Change in liver function as assessed by the Fibrosis-4 (FIB-4) index | Baseline, 6 months after enrollment
  The FIB-4 score consists of 4 variables including age,aspartate aminotransferase(AST), ALT, and platelets and evaluates the degree of fibrosis for patients suspected of or already diagnosed with hepatic fibrosis. Participants at low risk of advanced fibrosis have an index of less than 1.3 (age <65 years) or less than 2.0 (age ≥65 years); a score greater than 3.25 is suggestive of advanced fibrosis
Change in physical activity as assessed by the Actigraph GT9X accelerometers | Baseline, 6 months after enrollment
  Moderate-vigorous physical activity counts during the 7-day period will be calculated by summing moderate and vigorous activity counts and then applying a logarithmic transformation to address skew.
Change in physical activity as assessed by the International Physical Activity Questionnaire | Baseline, 6 months after enrollment
  This is a 27-item self-reported measure of physical activity. The result is reported categorically in one of three categories as follows: Low/inactive - do not meet the criteria for moderate or high activity levels, Moderate - meet 1 of the following: A) 3 or more days with at least 30 minutes of moderate-intensity activity or walking; B) 5 or more days with at least 30 minutes of moderate-intensity activity or walking; C) 5 or more days of any combination of walking, moderate-intensity, or vigorous intensity activities with at least 600 metabolic equivalent of task (MET)-minutes per week. [One MET is energy expenditure when at rest. For instance, 2 METs is twice the energy expended while at rest.] and high - meet 1 of the following: A: 3 or more days of vigorous-intensity activity and at least 1500 MET-minutes per week; B) 7 days of any combination of walking, moderate-intensity or vigorous intensity activities with at least 3000 MET-minutes per week.
Change in diet as assessed by the School Physical Activity & Nutrition (SPAN) survey - Healthy foods index | Baseline, 6 months after enrollment
  The School Physical Activity and Nutrition (SPAN) questionnaire is a brief self-administered measure of dietary intake. The healthy foods index will be reported, and total score ranges from 0-50, with a higher score indicating more frequent intake of healthy foods.
Change in diet as assessed by the School Physical Activity & Nutrition (SPAN) survey - Unhealthy foods index | Baseline, 6 months after enrollment
  The School Physical Activity and Nutrition (SPAN) questionnaire is a brief self-administered measure of dietary intake. The unhealthy foods index will be reported, and total score ranges from 0-45, with a higher score indicating more frequent intake of unhealthy foods.
Change in alcohol use as assessed by the alcohol use disorders identification test (AUDITC) | Baseline, 6 months after enrollment
  alcohol use disorders identification test (AUDITC) is a 3 item measure and will give a general idea of how often participants are drinking alcohol and in what quantities
Change in social support for physical activity as assessed by the Social Support for Exercise scales | Baseline, 6 months after enrollment
  This scale has 13 items, each is scored from 1(none)-5(very often) and 8(does not apply), higher number indicating better social support
Change in social support for diet as assessed by the Social Support for Diet scales | Baseline, 6 months after enrollment
  This scale has 10 items each is scored from 1(none)-5(very often) and 8(does not apply)
Change in participant illness perception as assessed by the brief Illness Perception Questionnaire | Baseline, 6 months after enrollment
  This is a 9 item questionnaire. The first 8 questions are scored from 0-10 and the 9th question will ask the subject to list in rank-order the three most important factors that they believe caused their illness.
Change in perceived severity | Baseline, 6 months after enrollment
  Perceived severity will be measured with 2 adapted items that assess to what extent they believe fatty liver disease is a severe health problem and to what extent do they consider complications for fatty liver to be severe health problems. Participants respond on a scale of 1-5, with a higher number indicating a perception that NAFLD is extremely severe.
Change in Perceived treatment efficacy | Baseline, 6 months after enrollment
  Perceived treatment efficacy will be assessed with 8 items, also adapted from Glasgow et al.that assess the importance of four protective factors (weight loss, eating healthy, avoiding sweets, and physical activity) and the likeliness of those factors to prevent future complications from fatty liver disease. Participants respond on a scale of 1-5, with a higher number indicating higher confidence in NAFLD treatment .
Change in Stress as assessed by the 4 items Perceived Stress Scale | Baseline, 6 months after enrollment
  Each of the 4 items is scored form (never)-4(very often) with a highest score of 16,indicating more stress
Change in Depression as assessed by the 10-item Center for Epidemiologic Studies Depression Scale (CESD-10) | Baseline, 6 months after enrollment
  This scale consists of 10 questions each one is scored form rarely or none of the time to all of the time.The total score is calculated by finding the sum of 10 items. Any score equal to or above 10 is considered depressed.
Change in Anxiety as assessed by the 7-item Generalized Anxiety Disorder (GAD-7) questionnaire. | Baseline, 6 months after enrollment
  This scale consists of 7 questions and each is scored form 0(not at all) to 3(nearly every day) for a maximum score of 21, a higher score indicating more anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Natalia I Heredia, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No